CLINICAL TRIAL: NCT01656798
Title: An Open-Label, Randomized, Single-Dose, 2-Way Crossover Study In Healthy Subjects Assessing The Pharmacokinetics And Safety Of Powder For Oral Suspension Of Sildenafil Citrate Administered Under Fasted And Fed Conditions
Brief Title: Food Effect Study For New Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A1481313
Record Dates: First submitted 2012-08-01; First posted 2012-08-03 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Healthy
MeSH Terms: interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- fasted condition (Experimental)
  Interventions: Drug: sildenafil citrate
- fec condition (Experimental)
  Interventions: Drug: sildenafil citrate

INTERVENTIONS:
Drug: sildenafil citrate — 2 mL of POS formulation of sildenafil citrate 10 mg/mL (equivalent to 20 mg dose), single dose
  Arms: fasted condition
Drug: sildenafil citrate — 2 mL of POS formulation of sildenafil citrate 10 mg/mL (equivalent to 20 mg dose), single dose
  Arms: fec condition

SUMMARY:
The main objective of this study is to estimate the effect of food on sildenafil pharmacokinetics after administration of Powder Oral Suspension (POS) formulation of sildenafil citrate.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 21 and 55 years
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >45 kg (99 lbs).

Exclusion Criteria:

* Baseline orthostatic hypotension defined as a ≥20 mm Hg reduction in systolic blood pressure (SBP), a ≥10 mm Hg reduction in diastolic blood pressure (DBP) or the development of significant postural symptoms (dizziness, lightheadedness, vertigo) when going from the supine to standing position.
* Subjects who are currently prescribed and/or taking nitrates or nitric oxide donors in any form on either a regular or intermittent basis.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of sildenafil | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12,14 hours post-dose
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] of sildenafil | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12,14 hours post-dose

SECONDARY OUTCOMES:
Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast) of sildenafil | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12,14 hours post-dose
Time to Reach Maximum Observed Plasma Concentration (Tmax)of sildenafil | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12,14 hours post-dose
Plasma Decay Half-Life (t1/2) of sildenafil | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12,14 hours post-dose
Maximum Observed Plasma Concentration (Cmax) of UK-103,320 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12,14 hours post-dose
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] of UK-103,320 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12,14 hours post-dose
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of UK-103,320 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12,14 hours post-dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) of UK-103,320 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12,14 hours post-dose
Plasma Decay Half-Life (t1/2) of UK-103,320 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12,14 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481313&StudyName=Food%20Effect%20Study%20For%20New%20Formulation